CLINICAL TRIAL: NCT07161102
Title: The Use of Foot Reflexology in Alleviating Anxiety Symptoms: A Randomized Clinical Trial
Brief Title: Effect of Foot Reflexology on Anxiety
Acronym: REFLEX-ANS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos Germano Dias Santos (Other)
Responsible Party: Sponsor-Investigator, Carlos Germano Dias Santos, Principal Investigator, Centro Universitário Maurício de Nassau
Organization: Centro Universitário Maurício de Nassau (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNINASSAU-REFLEXO-GERMANO-2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Reflexology; Foot Reflexology; Complementary Therapies; Integrative Health; POMS; BAI; Sham Massage
MeSH Terms: conditions — Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Reflexology (Experimental): Participants will receive 10 foot reflexology sessions, administered twice a week, each lasting approximately 30 minutes. The technique will be performed on specific reflexology points on the feet, according to protocols described in the scientific literature, aiming to reduce anxiety symptoms.
  Interventions: Other: Reflexology
- Sham Reflexology (Sham Comparator): Participants will receive 10 simulated intervention sessions, administered twice a week, each lasting approximately 30 minutes. The technique will consist of light, superficial touches to the feet, without stimulating reflexology points, with the aim of simulating the intervention without specific therapeutic effects.
  Interventions: Other: Sham Reflexology

INTERVENTIONS:
Other: Reflexology — A complementary technique that involves applying pressure to reflexology points on the feet. In this study, foot reflexology will be applied in 10 sessions, twice a week, for 30 minutes, aiming to reduce anxiety symptoms.
  Arms: Foot Reflexology
Other: Sham Reflexology — A simulated procedure consisting of superficial and random maneuvers on the feet, without stimulation of specific reflexology points. Ten sessions will be conducted twice a week, each lasting 30 minutes, for placebo control purposes.
  Arms: Sham Reflexology

SUMMARY:
This randomized, sham-controlled, parallel, double-blind clinical trial investigates the effects of foot reflexology on anxiety and well-being in adults with anxiety disorders. Participants are randomized (1:1) to receive either standardized foot reflexology or sham massage for 10 sessions (twice per week, 5 weeks). The primary outcome is the change in Beck Anxiety Inventory (BAI) score from baseline to the 10th session. Secondary outcomes include BAI score at 30-day follow-up, relaxation and well-being assessed immediately after each session with the Profile of Mood States (POMS - Brazilian version, Tension-Anxiety subscale), and incidence of adverse events. It is hypothesized that foot reflexology will result in a greater reduction of anxiety symptoms compared to sham massage.

DETAILED DESCRIPTION:
Participants aged 18-60 years with a clinical diagnosis of anxiety (DSM-5) are recruited and randomized 1:1 into two groups:

Experimental: standardized foot reflexology protocol targeting reflex points (solar plexus, CNS, pituitary, heart, diaphragm).

Sham comparator: foot manipulation and mobilization (sliding, flexion-extension, rotation, traction) without stimulation of reflex points.

Both interventions last approximately 15 minutes per session, 10 sessions total (twice per week for 5 weeks).

Assessments:

BAI at baseline, after 5 sessions, after 10 sessions, and 30-day follow-up. POMS (Tension-Anxiety subscale) immediately after each session (sessions 1-10). Checklist for adverse events (e.g., redness, pain, tingling, transient discomfort).

Blinding: Participants, care providers, outcome assessors, and statisticians are blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Clinical diagnosis of anxiety disorder confirmed by a healthcare professional (physician or psychologist).
* Score ≥ 11 on the Beck Anxiety Inventory (BAI) in the initial assessment.
* Availability to participate in the 10 proposed sessions.
* Signed informed consent.

Exclusion Criteria:

* Current use of benzodiazepines, antidepressants, or other psychotropic medications initiated less than 3 months ago.
* Associated diagnosis of psychotic disorder, bipolar disorder, or active suicidal ideation.
* Presence of serious or decompensated medical conditions (e.g., severe cardiovascular disease, uncontrolled epilepsy).
* Simultaneous participation in other complementary therapies (e.g., acupuncture, auriculotherapy, yoga, Reiki) during the study period.
* Pregnant or lactating women.
* Individuals with foot injuries, infections, or diseases that prevent foot reflexology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of Anxiety Symptoms (BAI) | Baseline, after 5 sessions and after 10 sessions (approximately 5 weeks).
  Anxiety symptom variation was assessed using the Beck Anxiety Inventory (BAI), a validated and widely used scale for measuring the intensity of anxiety symptoms. The total score ranges from 0 to 63, with higher scores indicating greater anxiety. The analysis will compare the scores obtained in the first session (baseline), the fifth session, and the tenth intervention session.

SECONDARY OUTCOMES:
Reduction of tension-anxiety levels (Profile of Mood States - POMS, reduced version) | Baseline, after 5 sessions (approximately 2.5 weeks), and after 10 sessions (approximately 5 weeks).
  Assessment of subjective perception of relaxation and psychological well-being using the Tension-Anxiety subscale of the Profile of Mood States (POMS) - Reduced Version, validated for Portuguese. Scores range from 0 to 36, with higher scores indicating greater tension and anxiety and lower scores indicating greater relaxation and well-being.
Recording of adverse effects related to the intervention | Throughout the intervention period (10 sessions - approximately 5 weeks).
  Systematic monitoring and recording of any adverse effects reported during or after foot reflexology or sham reflexology sessions, including pain, discomfort, or unexpected reactions. Outcomes will be categorized by frequency (number of participants affected) and intensity (mild, moderate, severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário Mauricio de Nassau, Vitória da Conquista, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT07161102/Prot_001.pdf